CLINICAL TRIAL: NCT03374605
Title: Modulating Context Generalization Through Transcranial Direct Current Stimulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This small mechanistic pilot study was ended prior to first enrollment after considering factors related to feasibility (e.g., available time and resources).
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1705-002
Record Dates: First submitted 2017-12-12; First posted 2017-12-15 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Anxiety and Fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental)
  Interventions: Device: active tDCS
- Sham tDCS (Sham Comparator)
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: active tDCS — 15 minutes of active (2mA) high definition tDCS will be applied to the participant's skull. The anodal electrode will be placed over 10-20 EEG coordinate AF7 and cathodal electrode over coordinate Fz.
  Arms: Active tDCS
Device: sham tDCS — 15 minutes of sham high definition tDCS will be applied to the participant's skull. The anodal electrode will be placed over 10-20 EEG coordinate AF7 and cathodal electrode over coordinate Fz.
  Arms: Sham tDCS

SUMMARY:
Behavioral adaptation is particularly relevant to anxiety and related disorders, where exposure-based therapies rely on such adaptation as part of behavior therapy.. However, while initial fear reactions generalize easily across contexts, subsequent adaption of behavior through learning is context-specific. The primary goal of this study is to investigate whether transcranial direct current stimulation (tDCS) can be used to acutely impact generalization of subsequent learning across contexts in an experimental paradigm. As part of this study, participants will complete a clinical interview and questionnaires, as well as a computer task asking them to make choices between stimuli on the screen and during which they may or may not receive tDCS.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of an anxiety or related disorder, (defined as panic disorder, social anxiety disorder, generalized anxiety disorder, obsessive-compulsive disorder, and/or post-traumatic stress disorder);
2. aged 18-55;
3. ability to speak, read, write, and understand English sufficiently well to complete study procedures and provide informed consent;
4. Stable psychiatric medication use for at least 6 weeks.

Exclusion Criteria:

1. Lifetime history of psychotic symptoms or bipolar disorder,
2. Current substance use disorder;
3. Acute suicidality or homicidality,
4. Significant neurological disorder,
5. Any problems that would interfere with study participation, significant or unstable medical disorders and tDCS-related contraindications (e.g., implanted metallic substances, pregnancy, holes in the skull, skin abnormalities under stimulation sites).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-02 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Relative frequency of selection of task-specific stimuli | 1 hour (measurement occurs 1 time only)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Garnaat, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No